CLINICAL TRIAL: NCT02345057
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate Efficacy and Safety of CS-3150 in Japanese Subjects With Type 2 Diabetes Mellitus and Microalbuminuria
Brief Title: A Study to Evaluate Efficacy and Safety of CS-3150 in Japanese Type 2 Diabetic Subjects With Microalbuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS3150-B-J204
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2016-09

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy; mineralocorticoid receptor antagonist; CS-3150; Japanese
MeSH Terms: conditions — Diabetic Nephropathies | interventions — esaxerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CS-3150 0.625 mg (Experimental): One CS-3150 0.625 mg tablet and one placebo tablet to match CS-3150 tablet administered orally, once daily after breakfast.
  Interventions: Drug: CS-3150; Drug: placebo
- CS-3150 1.25 mg (Experimental): Two CS-3150 0.625 mg tablets administered orally, once daily after breakfast.
  Interventions: Drug: CS-3150
- CS-3150 2.5 mg (Experimental): One CS-3150 2.5 mg tablet and one placebo tablet to match CS-3150 tablet administered orally, once daily after breakfast.
  Interventions: Drug: CS-3150; Drug: placebo
- CS-3150 5.0 mg (Experimental): Two CS-3150 2.5 mg tablets administered orally, once daily after breakfast
  Interventions: Drug: CS-3150
- Placebo (Placebo Comparator): Two placebo tablets to match CS-3150 tablet, administered orally, once daily after breakfast.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CS-3150
  Arms: CS-3150 0.625 mg; CS-3150 1.25 mg; CS-3150 2.5 mg; CS-3150 5.0 mg
Drug: placebo
  Arms: CS-3150 0.625 mg; CS-3150 2.5 mg; Placebo

SUMMARY:
This study is a randomized, placebo-controlled, double-blind, multi-center study to evaluate efficacy and safety of different doses of CS-3150 compared to placebo in Japanese Type 2 Diabetes Mellitus and Microalbuminuria.

The Primary endpoint is the change from baseline in urinary albumin to creatine ratio (UACR).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus
* Male or female subjects aged 20 years or older at informed consent
* Subjects with urinary albumin to creatine ratio (UACR) ≥ 45 mg/g Cr and < 300 mg/g Cr
* Estimated glomerular filtration rate by creatinine (eGFRcreat) ≥ 30 mL/min/1.73 m^2
* Subjects treated with angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) for at least 3 months prior to treatment period

Exclusion Criteria:

* Type 1 diabetes
* HbA1c (NGSP) >=8.4%
* Secondary glucose intolerance
* Subjects diagnosed with non-diabetic nephropathy
* Nephrotic syndrome
* Secondary hypertension or malignant hypertension
* Serum potassium level in any of the following categories: For subjects with eGFRcreat of ≥ 45 mL/min/1.73 m^2, serum potassium level of < 3.5 mEq/L or ≥ 5.1 mEq/L; For subjects with eGFRcreat of ≥ 30 mL/min/1.73 m^2 and < 45 mL/min/1.73 m^2, serum potassium level of < 3.5 mEq/L or ≥ 4.8 mEq/L

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urinary albumin to creatine ratio (UACR) | Baseline to end of Week 12

SECONDARY OUTCOMES:
Transition from microalbuminuria to normoalbuminuria | Baseline to end of Week 12
Change in renal function | Baseline to end of Week 12
Change in serum potassium | Baseline to end of Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Kumamoto, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592